CLINICAL TRIAL: NCT06704815
Title: Observational Cohort Study Evaluating the Effectiveness of an Educational Program (NGAYDAUTIEN) in Combination With Perindopril and Amlodipine Single-Pill Combination in Hypertensive Patients naïve of Antihypertensive Treatments.
Acronym: EDUHYPER
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-05985-004
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: observational; blood pressure; SBP; DBP; hypertension; HBP; HTA; Viacoram®; Perindopril arginine and Amlodipine; patient educational program
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Viacoram® plus educational program: naïve treatment hypertensive patients who will be initiated to Viacoram® plus an educational program
- other antihypertensive drugs (except Viacoram®): naïve treatment hypertensive patients who will be initiated to any antihypertensive drug (except single pill combination)

SUMMARY:
The primary objective is to assess the change of systolic blood pressure from baseline after a 6-month follow up for hypertensive patients initiating Viacoram® plus an educational program (NGAYDAUTIEN) in comparison to hypertensive patients initiating other antihypertensive drugs (except single pill combination).

ELIGIBILITY:
Inclusion Criteria:

1. Aged of at least 18 years (without upper limit of age)
2. Diagnosis of grade 1 or grade 2 hypertension
3. Naïve of treatment:

   * newly diagnosed hypertension and without treatment with antihypertensive effect for at least 3 months
   * previously diagnosed but without treatment with antihypertensive effect for at least 3 months
4. Patients follow-up within the scope of the current medical practice and in the same health centre during the 6-month period

Exclusion Criteria:

1. Previously attended to the Ngay Dau Tien educational program for HBP management
2. Plan to be hospitalized for other medical conditions during the next 6 months
3. Plan to move/relocate during 6-month follow-up
4. Have a severe disease (i.e. cirrhosis, end-stage renal disease …)
5. Are unlikely to cooperate in the study
6. Arm 1: patient having contra-indication to take Viacoram® according to SmPC
7. Arm 2: patient showing interest in attending NDT educational program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female who have a diagnosis of grade 1 or 2 hypertension and who initiate a new antihypertensive treatment
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
change of systolic blood pressure (measured in mmHg) from baseline after a 6-month follow up among the 2 arms | from baseline to 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Servier Affaires Médicales, Suresnes, France

IPD SHARING:
Plan to Share IPD: No